CLINICAL TRIAL: NCT02480959
Title: Functional Outcome of Surgical Treatment for Recurrent Patellar Instability: A Prospective Comparative Study Between Medial Retinacular Plication Versus Medial Patellofemoral Ligament Reconstruction
Brief Title: Medial Retinacular Plication Versus Medial Patellofemoral Ligament Reconstruction for Recurrent Patellar Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Rambam Health Care Campus (Other); Hadassah Medical Organization (Other); Assaf-Harofeh Medical Center (Other Government); Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0041-15-MMC
Record Dates: First submitted 2015-06-08; First posted 2015-06-25 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Patella, Familial Recurrent Dislocation Of
MeSH Terms: conditions — Patella, Familial Recurrent Dislocation Of | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medial plication (Other): Patient undergoing surgical treatment for recurrent patellar instability that includes medial retinacular plication
  Interventions: Procedure: Surgical treatment for recurrent patellar instability
- MPFL reconstruction (Other): Patient undergoing surgical treatment for recurrent patellar instability that includes medial patellofemoral ligament reconstruction using a tendon graft
  Interventions: Procedure: Surgical treatment for recurrent patellar instability

INTERVENTIONS:
Procedure: Surgical treatment for recurrent patellar instability — Either medial plication or MPFL reconstructuion surgery

SUMMARY:
The purpose of this study is to determine whether medial patellofemoral ligament reconstruction results in superior functional outcomes compared to medial retinacular plication surgery in cases of recurrent patellar instability.

DETAILED DESCRIPTION:
Patients with recurrent lateral patellar instability will be assigned to undergo one of two surgical approaches aimed to prevent recurrent patellar instability and result in improvement in function. One surgical approach will be medial retinacular plication with multiple stitches while the other surgical approach will include medial patellofemoral ligament reconstruction using a hamstring tendon graft. Prior to surgery, and then during follow-up after surgery as well as at the completion of minimum two years follow-up after surgery, patients will be asked to complete subjective functional questionaires that will rate their knee function, and to undergo detailed physical examination and objective functional tests that will quantify the success of surgery. The outcomes of the surgical treatment options will be compared to determine whether medial patellofemoral ligament reconstruction results in superior function and patient subjective satisfaction compared to medial retinacular plication only.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent lateral patellar instability has been described by the patient

Imaging criteria include:

* TT-TG distance (on CT or MRI) is between 10-20 mm
* Insall-Salvati Index is between 0.9 - 1.2
* Trochlea angle is lower than 145 degrees

Exclusion Criteria:

* Only a single event of lateral patellar instability occured

Imaging criteria include:

* TT-TG distance (on CT or MRI) is below 10 mm or above 20 mm
* Insall-Salvati Index is below 0.9 or above 1.2
* Trochlea angle is above 145 degrees
* Other concomitant intra-articular patholgies, injuries, and surgeries, besides the patella instability, with were recorded at the lower limbs and did not uneventfuly healed, and as a result cause dysfunction of the lower limbs
* Significant ligamentous injuries of the knees, including cruciate and collateral injuries, as well as meniscal injuries that interfere with function

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Kujala knee outcome score | Between two and five years after surgery
  A validated international outcome score that evaluates knee functional outcome in relation to patellofemoral symptoms

SECONDARY OUTCOMES:
International Knee Documentation Committee subjective outcome score | Between two and five years after surgery
  A validated international outcome score that evaluates general knee functional outcome
Tenger activity level score | Between two and five years after surgery
  A validated international outcome score that evaluates highest level of sports activity
Marx activity level score | Between two and five years after surgery
  A validated international outcome score that evaluates highest level of sports activity
Visual Analogue Scale | Between two and five years after surgery
  A validated international scale that evaluates level of pain
Single hop test | Between two and five years after surgery
  Evaluates limb asymmetry index between operated and nonoperated limbs during a single legged hop for distance
Side-to-side hop test | Between two and five years after surgery
  Evaluates limb asymmetry index between operated and nonoperated limbs performing side to side repetaed hops during 30 seconds
Patellar apprehension test | Between two and five years after surgery
  Evaluates normal patellar tracking and patient's feeling of subjective comfort while the examiner apply a provocative force that translates the patella lateraly
Infectious event of the operated knee documented by number of events that required antibiotics treatment with or without joint lavage | Immediately after surgery, for the duration of hospital stay, and until expected time of 1 month
  Infection of the surgical site as a severe complication of surgery, requirng antibiotics with or without joint lavage

CONTACTS AND LOCATIONS:
Overall Officials: IFTACH HETSRONI, M.D., Principal Investigator — Meir Medical Center; DROR LINDNER, M.D., Principal Investigator — Assaf-Harofeh Medical Center; IDAN ILSAR, M.D., Principal Investigator — Hadassah Medical Organization; MAZEN FALAH, M.D., Principal Investigator — Rambam Health Care Campus; NASSIM ALKRINAWI, M.D., Principal Investigator — Soroka University Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel